CLINICAL TRIAL: NCT04474613
Title: Use of Liquid Biopsy to Reduce Time to Treatment for Patients With Advanced Nonsquamous Non-small Cell Lung Cancer Diagnosed at Outside Sites
Brief Title: Liquid Biopsy to Reduce Time to Treatment for Advanced Nonsquamous NSCLC Diagnosed at Outside Sites
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE1520
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Liquid Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liquid biopsy (Experimental): A liquid biopsy is a test will be done on a sample of blood to look for cancer cells
  Interventions: Diagnostic Test: Liquid biopsy

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — Liquid biopsy done on a blood draw, taking approximately 7 days

SUMMARY:
The purpose of this study is to determine if liquid biopsies will reduce time to begin treatment in participants with non-small cell lung cancer (NSCLC). A liquid biopsy is a test done on a sample of blood to look for cancer cells.

DETAILED DESCRIPTION:
Referred patients with newly diagnosed NSCLC who have not had genetic testing for targetable mutations will be considered for this study. The primary objective of this prospective study is to examine if using liquid biopsy can reduce time to treatment (TTT) in external participants with NSCLC. Secondary objectives examined will include time to actionable genetic testing results (ctDNA or tissue), rate of actionable biomarker discovery, and rate of appropriate guideline-directed therapy based upon testing results.

A liquid biopsy is a test done on a sample of blood to look for cancer cells. A traditional biopsy, which requires tissue to be removed from the body, takes 14 days to be tested. A liquid biopsy takes 7 days which significantly shortens the TTT for those diagnosed with NSCLC. By studying this, doctors may be better able to determine if this will be beneficial and result in less time taken to treat cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants with newly diagnosed, advanced nonsquamous NSCLC referred to the Cleveland Clinic Taussig Cancer Center from outside centers without prior testing results available for targetable genetic alterations
* Plan to receive systemic therapy at the Cleveland Clinic, OR plan to receive systemic therapy at an outside site while maintaining either intermittent follow up at Cleveland Clinic or with electronic health record access through Care Everywhere.

Exclusion Criteria:

* Prior therapy for this diagnosis of NSCLC
* Prior adequate molecular testing done for the current diagnosis of NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
TTT measured in days | An average of 30 days
  TTT measured in days - TTT will be summarized using mean, SD, and range. One sample t-test will be used to compare observed TTT against the null (30 days).

SECONDARY OUTCOMES:
Time to actionable genetic testing results | An average of 30 days
  Time to actionable genetic testing results (ctDNA or tissue). Negative results with ctDNA testing will still require tissue confirmation, while positive results will be considered actionable without further testing.
Rate of actionable biomarker discovery | An average of 30 days
  Rate of actionable biomarker discovery, defined as the percentage of tested patients who have a detected genetic marker that is associated with either 1) an FDA-approved targeted treatment or 2) a targeted treatment available through a clinical trial.
Rate of appropriate guideline-directed therapy based upon testing results | An average of 30 days
  Rate of appropriate guideline-directed therapy based upon testing results

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Pennell, MD, PhD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies the publication
Supporting Information: Study Protocol, ICF
Time Frame: Shortly after completion of the study which is to take approximately one year